CLINICAL TRIAL: NCT00349180
Title: Multicenter, Randomized, Double-Blind Study to Evaluate the Efficacy and Safety of Enoxaparin Sodium（RP54563）20mg qd and 20mg Bid for 14 Days in Patients With Total Hip Replacement
Brief Title: Total Hip Replacement Study With XRP4563 (Enoxaparin Sodium)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC6770
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Total Hip Replacement; Enoxaparin
MeSH Terms: interventions — enoxaparin sodium

INTERVENTIONS:
Drug: Enoxaparin sodium

SUMMARY:
This study is performed to confirm the optimal dose for THR (total hip replacement).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective primary THR (total hip replacement) surgery

Exclusion Criteria:

* Patient with risk of clinical significant bleeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156
Dates: Start 2006-06

PRIMARY OUTCOMES:
Incidence of VTE

SECONDARY OUTCOMES:
Incidence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro IKEDA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan